CLINICAL TRIAL: NCT04872140
Title: Effect of Low-phytate Pea Powder With High Iron Bioavailability on Iron Status of Female Runners
Brief Title: Effect of Iron-fortified Pea Powder on Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1207
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Participants are being randomized to three groups for the 8-week intervention:
  1. Pea power with high iron bio-availability
  2. Regular pea powder
  3. Placebo (maltodextrin)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The powder supplements are being administered in a blinded manner. An individual who is separate from the rest of the research team will generate the allocation schedule and prepare the supplement packages so that participants, investigators, and outcome assessors are blinded. Statistical analysis will be blinded by coding of groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pea power with high iron bio-availability (Experimental): Pea powder with low phytate levels to increase iron bio-availability (7mg iron per day)
  Interventions: Dietary Supplement: Low phytate pea powder
- Pea powder (Active Comparator): Pea powder with normal phytate levels (7mg iron per day)
  Interventions: Dietary Supplement: Regular pea powder
- Placebo (Placebo Comparator): Placebo (maltodextrin) powder (0g iron per day)
  Interventions: Dietary Supplement: Placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Low phytate pea powder — Exercise performance with low phytate pea powder
  Arms: Pea power with high iron bio-availability
Dietary Supplement: Regular pea powder — Exercise performance with regular pea powder
  Arms: Pea powder
Dietary Supplement: Placebo (maltodextrin) — Exercise performance with placebo (maltodextrin)
  Arms: Placebo

SUMMARY:
Female endurance athletes are susceptible to iron deficiency and this can impact their exercise performance. This study assesses the impact of an pea protein supplement with high iron bio-availability on iron status and exercise performance.

DETAILED DESCRIPTION:
Female endurance athletes are susceptible to iron deficiency due to poor iron intake from diets or possibly because of destruction of red blood cells during foot-strike hemolysis. This study will evaluate the impact of 8-weeks of iron supplementation through consumption of a pea-protein power that has high iron bio-availability due to low phytate levels. This will be compared to consumption of regular iron protein powder and maltodextrin placebo by randomizing participants to three groups. Participants will be assessed at baseline and after 8 weeks of supplementation for exercise performance (maximal aerobic capacity and a 5 km time trial running test), blood levels of ferritin and hemoglobin, and body composition (fat mass and lean tissue mass).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Regularly participate in aerobic endurance training

Exclusion Criteria:

* Any contra-indications to exercise testing as determined with the "Get Active Questionnaire"

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ferritin levels | Up to 8 weeks
  blood ferritin levels

SECONDARY OUTCOMES:
Change from baseline in maximal aerobic capacity | Up to 8 weeks
  Maximal aerobic capacity (mL/kg/min) measured on a treadmill
Change from baseline in exercise time trial performance | Up to 8 weeks
  Time (minutes) to complete 5 km running on a treadmill
Change from baseline in hemoglobin levels | Up to 8 weeks
  Blood hemoglobin concentration
Change from baseline in lean tissue mass | Up to 8 weeks
  Lean tissue mass (kg) measured with dual energy X-ray absorptiometry
Change from baseline in fat mass | Up to 8 weeks
  Fat mass (kg) measured with dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw KA, Chilibeck PD, Lindsay DL, Warkentin TD, Ko J, Zello GA. Low phytic acid pea supplementation as an approach to combating iron deficiency in female runners: A randomized control trial. Nutr Health. 2025 Mar;31(1):293-301. doi: 10.1177/02601060231181605. Epub 2023 Jun 8. PMID 37291968